CLINICAL TRIAL: NCT01710085
Title: Diagnostic Value of Diffusion Weighted Imaging in Detection of Recurrent Disease in Cervical and Endometrial Cancer Treated With Curative Surgery
Brief Title: Value of Diffusion Weighted Magnetic Resonance Imaging in Detection of Recurrent Disease in Surgically Treated Cervical and Endometrial Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Kadir Hacikurt, Dr. Kadir Hacıkurt, Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: KUAP(T)-2012/39
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Cervical Cancer; Endometrial Cancer
Keywords: Diffusion weighted MRI; Curative surgery; Recurrence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Recurrence | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diffusion weighted imaging, Recurrence (Experimental)
  Interventions: Device: Diffusion weighted MRI (DW- MRI)- Philips Achieva 3.0T X, Netherlands, 2011

INTERVENTIONS:
Device: Diffusion weighted MRI (DW- MRI)- Philips Achieva 3.0T X, Netherlands, 2011 — Recurrence in cervical and endometrial cancer patients who were treated with curative surgery is routinely investigated by MRI examination. MRI is diagnostic technique not requiring ionizing radiation and is based on magnetic fields.

SUMMARY:
Endometrial and cervical cancers are one of the most common malignancies seen in females. Identification of recurrent disease in early phases of treatment carries a primary importance on the outcome of patients. Diffusion-weighted magnetic resonance imaging (DWI) is a new technique recently started to be performed in body imaging and has potential ability to detect recurrent disease. The aim of this study is to investigate the diagnostic impact of DWI in detection of recurrent disease in patients treated with curative surgery in endometrial and cervical cancer.

DETAILED DESCRIPTION:
Endometrial and cervical cancers are one of the most common malignancies seen in female genital tract. Although, surgical resection is the treatment of choice for both, adjuvant or neo-adjuvant chemotherapy or radiotherapy and curative radiotherapy are alternative treatment options depending on the stage.

Identification of recurrent disease in early phases carries a primary importance on the prognosis.

Diffusion-weighted MRI (DWI), a new technique recently started to be performed in body imaging has potential ability to distinguish recurrent disease from normal tissue or fibrosis. Our aim in this study is to investigate the diagnostic impact of DWI in detection of recurrence rate in patients treated with curative surgery in endometrial and cervical cancer.

All patients who had curative surgery due to endometrial or cervical cancer will be included to the study. Patients will be examined with DWI in addition to routine sequences including contrast enhanced dynamic studies. The sensitivity, specificity, accuracy as well as positive and negative predictive values of the study will be investigated from the data derived from DWI studies and will be correlated with data obtained by conventional radiologic, nuclear imaging studies including PET-CT, as well as pathologic verifications during follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of cervical or endometrial cancer.
* Patients treated with curative surgery (hysterectomy)will be involved on a voluntary basis.

Exclusion Criteria:

* Contraindications for MRI examination (cardiac pacemakers, metallic objects, cochlear implants, claustrophobic patients)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Investigation of the diagnostic value of DWI in detection of recurrence rate in patients treated with curative surgery in endometrial and cervical cancer. | 18 months
  Postoperative recurrent disease is usually investigated with physical examination, ultrasonography, computed tomography (CT), conventional magnetic resonance imaging (MRI) and positron emission tomography-computed tomography (PET-CT) with different sensitivity and specificities. However, radiologists experience difficulty in detection of small recurrent active tumors with anatomically-based radiologic modalities like CT or conventional MRI in patients treated with hysterectomy. Furthermore, effects of adjuvant therapies or fibrosis developed following surgery could mask or even mimic the recurrent tumor. Our aim in this study is to investigate the diagnostic impact of DWI in detection of recurrence rate in patients treated with curative surgery in endometrial and cervical cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Gürsel Savcı, Prof., Study Director — Uludag University; Kadir Hacıkurt, Dr., Principal Investigator — Uludag University
Locations (1):
- Uludağ Üniversitesi, Bursa, Turkey (Türkiye)